CLINICAL TRIAL: NCT06252181
Title: Pain and Hemodynamics in Peripheral Arterial Disease: Response to Pulsed Electromagnetic Treatment in Elderly
Brief Title: Pain and Hemodynamics in Peripheral Arterial Disease: Response to Pulsed Electromagnetic Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Hagar Ahmed El-Hadidy, lecturer of physical therapy for Internal Medicine and Geriatrics, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004285
Record Dates: First submitted 2024-02-02; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): group of peripheral arterial disease elderly (n=20) that take their medications and will receive 3 sessions per weeks of 8-week electromagnetic one-hour therapy and one hour elliptical exercise (exercise will be applied 3 times per the week for eight week)
  Interventions: Other: electromagnetic pulsed therapy
- group number 2 (Active Comparator): patients (20 elderly) with peripheral arterial disease who take their medications will receive one hour elliptical exercise ( exercise will be applied 3 times per the week for eight week)
  Interventions: Other: elliptical exercise

INTERVENTIONS:
Other: electromagnetic pulsed therapy — patients (20 elderly) with peripheral arterial disease who take their medications will receive one hour elliptical exercise ( exercise will be applied 3 times per the week for eight week) and 3 sessions per weeks of 8-week electromagnetic one-hour pulsed therapy
  Arms: group number 1
Other: elliptical exercise — patients (20 elderly) with peripheral arterial disease who take their medications will receive one hour elliptical exercise (n=20 patients, exercise will be applied 3 times per the week for eight week)
  Arms: group number 2

SUMMARY:
patients with peripheral arterial disease are recommended to perform all exercise forms including elliptical type. electromagnetic treatment addition to exercise may increase benefits of this exercise

DETAILED DESCRIPTION:
patients (40 elderly) with peripheral arterial disease who take their medications will be divided to older patients group that receive one hour elliptical exercise (n=20 patients, exercise will be applied 3 times per the week for eight week) and a group (n=20) that receive 3 sessions per weeks of 8-week electromagnetic one-hour therapy and one hour elliptical exercise (exercise will be applied 3 times per the week for eight week)

ELIGIBILITY:
Inclusion Criteria:

* older patients
* peripheral arterial disease patients

Exclusion Criteria:

* cardiac elders
* respiratory elders
* renal elders

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
ankle brachial index | It will be measured after 8 weeks
  it is an vascular index used in assessment of peripheral arterial disease progression

SECONDARY OUTCOMES:
posterior tibial artery diameter | It will be measured after 8 weeks
  increase in vascular diameter of vessel denotes improved arterial disease
claudication pain time | It will be measured after 8 weeks
  the starting onset time of pain appearance during treadmill test
claudication pain distance | It will be measured after 8 weeks
  the distance at which onset of pain appeared during treadmill test
Modified walking impairment questionnaire | It will be measured after 8 weeks
  it assess degree of walking impairment in vascular disease patients
six minute walking test (pain free distance) | It will be measured after 8 weeks
  pain free distance walked during six minute walking test will be calculated
six minute walking test (total walked distance) | it will be measured after 8 weeks
  total distance walked during six minute walking test will be calculated
intermittent claudication questionnaire | it will be measured after 8 weeks
  it will assess health-related quality of life concerning the issue of intermittent claudication
short form 36 health questionnaire | it will be measured after 8 weeks
  it will assess general quality of life in the patients
Short physical performance battery | it will be measured after 8 weeks
  total score or points will be assessed from this physical performance test

CONTACTS AND LOCATIONS:
Overall Officials: hagar El-Hadidy, lecturer, Principal Investigator — Ahram Canadian University
Locations (1):
- Ahram canadian university, Giza, Egypt